CLINICAL TRIAL: NCT05459142
Title: Safety and Acceptability of Telemedicine Medical Abortion Service Using the "No-test" Protocol in Azerbaijan.
Brief Title: Telemedicine Medical Abortion Service Using the "No-test" Protocol in Azerbaijan.
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Collaborators: Scientific Research Institute of Obstetrics and Gynecology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1057
Record Dates: First submitted 2022-07-12; First posted 2022-07-14 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2022-07

CONDITIONS: Pregnancy Related
Keywords: Telemedicine; Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Medical Abortion — Medical Abortion

SUMMARY:
The goal of this study is to pilot and evaluate a telemedicine medical abortion service delivery that allows remote communication between the woman and provider and limits medically unnecessary in-person visits to health or diagnostic centers.

DETAILED DESCRIPTION:
The goal of this study is to pilot and evaluate a telemedicine medical abortion (TMA) service delivery that allows remote communication between the woman and provider and limits medically unnecessary in-person visits to health or diagnostic centers. Providers will provide counseling by phone or video about pregnancy options and give detailed information about the medical abortion process, expected side effects, and where to seek additional care. The provider will then evaluate the woman's eligibility for TMA service by following the no-test protocol and discuss at-home follow-up using a symptom checklist and a high-sensitivity urine pregnancy test. If pre-treatment tests are needed, women will be referred to a nearby diagnostic center and test results will be forwarded to the study provider. Participants will receive medications by mail or courier service or pick them up at the pharmacy or study clinics, take medications as instructed, and complete at-home follow-ups as discussed with the provider.

ELIGIBILITY:
Inclusion Criteria:

* Is pregnant as determined by a pregnancy test or ultrasound (if obtained prior to contacting the study site)
* Has no contraindications to medical abortion
* Has access to a phone
* Is able to take mifepristone on or before 63 days of gestation

Exclusion Criteria:

* Medically ineligible for medical abortion
* Gestational age above 63 days based on LMP

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants who seek early first-trimester abortion at the participating study site and would like to receive telemedicine medical abortion services.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
The incidence rate of adverse events resulting from the remote provision of medical abortion | 6 weeks
  Adverse events such as regimen non-compliance or medically unnecessary interventions associated with remote provision of medical abortion.

SECONDARY OUTCOMES:
Satisfaction with remote provision of medical abortion | 6-weeks
  Satisfaction with remote provision of medical abortion measures by 5-point Likert scale. We will be using a 1-5 score system. 1 being very satisfied and 5 being very unsatisfied. A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific-Research Institute of Obstetrics and Gynecology, Baku, Azerbaijan

IPD SHARING:
Plan to Share IPD: No